CLINICAL TRIAL: NCT03467139
Title: The Effect of Abdominal Breathing Exercises on Pain, Sleep and Quality of Life in Patients With Adhesive Capsulitis
Brief Title: Breathing Exercises and Adhesive Capsulitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hasan Kalyoncu University (Other)
Responsible Party: Principal Investigator, YUSUF ŞİNASİ KIRMACI, Yusuf Şinasi Kırmacı,Principal Investigator,Physical Therapist, Hasan Kalyoncu University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: YusufKirmaci
Record Dates: First submitted 2018-02-09; First posted 2018-03-15 (Actual); Last update posted 2018-03-16 (Actual); Status verified 2018-03

CONDITIONS: Adhesive Capsulitis
Keywords: Adhesive Capsulitis; Breathing exercises; Pain; Sleep quality; Quality of life
MeSH Terms: conditions — Bursitis; Pain; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study Group (Experimental): Hotpack was applied for 15 min and TENS was applied for 15 min and ultrasonics for 5 min. Then scapular mobilization and passive stretching exercises were applied in 10 sets of 3 sets (flexion, abduction, internal and external rotation) to increase joint range of motion by physiotherapist. Then, abdominal breathing exercise training was given 3 times a week as 30 sets of 3 sets a week and the patients were treated for 8 weeks
  Interventions: Other: Abdominal breathing exercise
- Control Group (No Intervention): Hotpack was applied for 15 min and TENS was applied for 15 min and ultrasonics for 5 min. Then scapular mobilization and passive stretching exercises were applied for 8 weeks in 10 sets of 3 sets (flexion, abduction, internal and external rotation) to increase joint range of motion.

INTERVENTIONS:
Other: Abdominal breathing exercise — Deep Breathing Exercise
  Arms: Study Group

SUMMARY:
The purpose of this study was to determine the effects of abdominal breathing exercises on pain, sleep quality and quality of life with adhesive capsulitis patients. The 41 adhesive capsulitis patients, 29 women and 12 men aged between 40-65 years, had divided into two groups by simple random sampling. In the study group, abdominal breathing exercise training was applied to routine physiotherapy program, in the control group routine physiotherapy program was applied for 8 weeks. Individuals were assessed for lung function test, range of motion, pain, sleep quality and quality of life. First assesment were performed at the beginning of treatment, 2nd assesment were performed at the end of 8 th week.

DETAILED DESCRIPTION:
Pain in the early stages of adhesive capsulitis leads to many symptoms such as sleeping problems. Breathing exercises also began to take place among the applications towards pain. Abdominal respiration is considered the easiest method to reveal relaxation response. Slow breathing increases parasympathetic activity in the body and reduces sympathetic activity. This is the first and fundamental step of real healing. The reduction of pro-inflammatory markers with respiratory exercises suggests that respiratory exercises are effective in inflammation.

On study group; Hotpack was applied for 15 minutes and TENS was applied for 15 minutes and ultrasonics for 5 minutes. Then, scapular mobilization and passive stretching exercises were applied in 10 sets of 3 sets (flexion, abduction, internal and external rotation) to increase joint range of motion by physiotherapist. Then abdominal respiratory exercise training was given 3 times a week as 30 sets of 3 times a week and patients were treated for 8 weeks.

For the control group; Hotpack was applied for 15 min and TENS was applied for 15 min and ultrasonics for 5 min. Then scapular mobilization and passive stretching exercises were applied for 8 weeks in 10 sets of 3 sets (flexion, abduction, internal and external rotation) to increase joint range of motion by physiotherapist.

ELIGIBILITY:
Inclusion Criteria:

* Those who have received an adhesive capsulitis diagnosis,
* Those in the age range 40-65

Exclusion Criteria:

* Those who take medicine for pain,
* Those with a primary sleep problem,
* Those with respiratory system disease,
* Those with cognitive problems,
* Non-volunteer

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2017-03-24 (Actual); Primary Completion 2017-06-15 (Actual); Study Completion 2017-06-30 (Actual)

PRIMARY OUTCOMES:
Pain | Change from Baseline Pain at 8 weeks
  Visual Analog Scale-Min.score:0 Max.score:10.0 means no pain, 10 means unbearable pain.
Pain | Change from Baseline Pain at 8 weeks
  Shoulder Pain and Disability Index: It consists of 2 subtitles.First subtitle is pain, has 5 items. first subtitle: Min:0-Max:100. 0 means no pain in functional activities, and 100 means irresistible pain. Second subtitle is disability,has 8 items. Min. score is 0, Max score is 100. 0 means no disability in functional activities, 100 means disabile in functional activities. Total score changes 0-100. 0 shows best score, 100 shows worst score.
Sleep Quality | Change from Baseline Sleep Quality at 8 weeks
  Pittsburgh Sleep Quality Index-Min.score:0 Max.score:21. High total score indicates poor sleep quality.
Sleep Quality | Change from Baseline Sleep Quality at 8 weeks
  Epworth Sleepiness Scale.Min:0-Max:24.0 indicates no sleepiness, and 24 indicates max daytime sleepiness.
Quality of Life | Change from Baseline Quality of Life at 8 weeks
  SF-36:It consists of 36 items in total. It consists of 8 subtitles. (3 items), Energy (4 items), Mental Health (5 items), Social Function (2 items), Pain (2 items), General (10 items), Physical Role Strength Health Scale (8 items). The lower scales measure the health between 0 and 100, and 0 refers to the poor health status and 100 to the good health status.
Lung Function Test | Change from Baseline Lung Function at 8 weeks
  Lung Function Test

SECONDARY OUTCOMES:
Range of Motion | Change from Baseline Range of Motion at 8 weeks
  Universal Goniometer
Muscle Strength | Change from Baseline Muscle Strength at 8 weeks
  Manuel Muscle Strength Test

CONTACTS AND LOCATIONS:
Overall Officials: Hasan Kalyoncu University Health Sciences college, Principal Investigator — Hasan Kalyoncu University
Locations (1):
- Hasan Kalyoncu Unıversity, Gaziantep, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided